CLINICAL TRIAL: NCT04136171
Title: A Phase 3 Global, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Efficacy and Safety of ION-682884 in Patients With Transthyretin-Mediated Amyloid Cardiomyopathy (ATTR CM)
Brief Title: CARDIO-TTRansform: A Study to Evaluate the Efficacy and Safety of Eplontersen (Formerly Known as ION-682884, IONIS-TTR-LRx and AKCEA-TTR-LRx) in Participants With Transthyretin-Mediated Amyloid Cardiomyopathy (ATTR CM)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ION-682884-CS2; 2019-002835-27 (EudraCT Number); 2024-514434-20-00 (EU CTIS Number)
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Transthyretin-Mediated Amyloid Cardiomyopathy (ATTR CM)
Keywords: TTR; Amyloidosis; Cardiomyopathy
MeSH Terms: conditions — Amyloidosis; Cardiomyopathies | interventions — eplontersen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Eplontersen (Experimental): Eplontersen by subcutaneous injection once every 4 weeks
  Interventions: Drug: Eplontersen
- Placebo (Placebo Comparator): Eplontersen-matching placebo by subcutaneous injection once every 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eplontersen — Eplontersen by subcutaneous injection
  Other Names: ION-682884; IONIS-TTR-LRx
  Arms: Eplontersen
Drug: Placebo — Eplontersen-matching placebo by subcutaneous injection
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of eplontersen compared to placebo in participants with ATTR-CM receiving available standard of care (SoC).

DETAILED DESCRIPTION:
This is a multicenter, double-blind study in 1438 participants, who will be randomized to receive subcutaneous (SC) injections of either eplontersen or placebo once every 4 weeks. Participants will also receive daily supplemental doses of the recommended daily allowance of vitamin A.

ELIGIBILITY:
Inclusion Criteria:

* Females must be non-pregnant and non-lactating, and either surgically sterile or post-menopausal or abstinent. If engaged in sexual relations of child-bearing potential, agree to use 1 highly effective contraceptive method
* Males must be surgically sterile or, abstinent or, if engaged in sexual relations with a woman of child-bearing potential, the participant or the participant's non-pregnant female partner must be using a highly effective contraceptive method
* Amyloid deposits in cardiac or non-cardiac tissue confirmed by Congo Red (or equivalent) staining OR technetium scintigraphy (99mTc -3,3-diphosphono-1,2- propanodicarboxylic acid [DPD-Tc], 99m Tc-pyrophosphate [PYP-Tc], or 99m Tc-hydroxymethylene-diphosphonate [HMDP-Tc]) with Grade 2 or 3 cardiac uptake in the absence of abnormal light chains ratio, centrally confirmed
* End-diastolic interventricular septum thickness of > 12 millimeters (mm) on Screening echocardiogram
* New York Heart Association (NYHA) class I-III

Exclusion Criteria:

* Acute coronary syndrome, unstable angina, stroke, transient ischemic attack (TIA), coronary revascularization, cardiac device implantation, cardiac valve repair, or major surgery within 3 months of Screening
* Cardiomyopathy not primarily caused by ATTR-CM, for example, cardiomyopathy due to hypertension, valvular heart disease, or ischemic heart disease
* Monoclonal gammopathy of undetermined significance (MGUS) and/or alterations in immunoglobulin free light chain (FLC) ratio unless fat, bone marrow, or heart biopsy confirming the absence of light chain and the presence of TTR protein by mass spectrometry or immunoelectron microscopy. For participants with chronic kidney disease (CKD) and without presence of monoclonal protein in blood and urine, the acceptable FLC ratio is 0.26-2.25. Results different from that may be discussed with local hematologist, Investigator and Medical Monitor if the risks associated with the biopsy outweigh the benefits
* Prior liver or heart transplant, and/or Left Ventricular Assist Device (LVAD) or anticipated liver transplant or LVAD within 1 year after randomization
* Current or previous treatment with Tegsedi™ (inotersen) or Onpattro™ (patisiran) or other oligonucleotide or ribonucleic acid (RNA) therapeutic (including small interfering ribonucleic acid [siRNA]; does not apply to COVID-19 mitochondrial [mRNA] vaccinations)
* Current treatment with diflunisal, doxycycline, with or without ursodeoxycholic acid, and/or non-dihydropyridine calcium-channel blocker (e.g., verapamil, diltiazem). Participants receiving any of these agents must respect a wash-out period of 14 days before randomization.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1438 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Composite Outcome of Cardiovascular (CV) Mortality and Recurrent CV Clinical Events up to Week 140 | Baseline up to Week 140

SECONDARY OUTCOMES:
Change From Baseline in the 6-minute Walk Test (6MWT) Distance at Week 140 | Baseline to Week 140
  The 6MWT is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes. The 6MWT provides information regarding functional capacity, response to therapy and prognosis across a range of chronic cardiopulmonary conditions.
Change From Baseline in the Kansas City Cardiomyopathy Questionnaire (KCCQ) Scores at Week 140 | Baseline to Week 140
  The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a 23-item self-administered questionnaire developed to independently measure the participant's perception of their health status, which includes heart failure symptoms, impact on physical and social function, and how their heart failure impacts their quality of life (QOL) within a 2-week recall period.
  The KCCQ tool quantifies the following six (6) distinct domains and two (2) summary scores. KCCQ responses are provided along a rating scale continuum with equal spacing from worst to best, with a higher score equaling a better score.
Recurrent CV Clinical Events up to Week 140 | Baseline up to Week 140
All-Cause Mortality up to Week 160 | Baseline up to Week 160
All-Cause Mortality up to Week 140 | Baseline up to Week 140
Composite Outcome of Cardiovascular (CV) Mortality and Recurrent CV Clinical Events up to Week 140 in Subgroup of Patients Treated with Tafamidis at Baseline | Baseline up to Week 140
  To evaluate the effect of treatment with ION-682884 compared to placebo up to Week 140 on the composite endpoint of CV death and recurrent CV clinical events in patients with ATTR-CM on tafamidis at Baseline.
CV Mortality up to Week 160 | Baseline up to Week 160
CV Mortality up to Week 140 | Baseline up to Week 140

CONTACTS AND LOCATIONS:
Locations (142):
- United States (51):
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - Altman Clinical and Translational Research Institute Center for Clinical Research, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, San Francisco (UCSF) - Medical Center, San Francisco, California
  - Stanford Hospital, Stanford, California
  - University of Colorado Hospital - Anschutz Medical Campus, Aurora, Colorado
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - The George Washington Medical Faculty Associates - Foggy Bottom North Pavilion, Washington D.C., District of Columbia
  - Cleveland Clinic Florida, Weston, Florida
  - Emory Heart and Vascular Center - Emory Clifton Campus, Atlanta, Georgia
  - Piedmont Heart of Fayetteville, Fayetteville, Georgia
  - Northwestern University, Chicago, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana University Health, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Louisiana State University Health Sciences Center, New Orleans, Louisiana
  - Tulane University Heart and Vascular Institute, New Orleans, Louisiana
  - Ochsner Health System, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - New York University Langone Cardiology Associates, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Weill Cornell Medicine Cardiology, New York, New York
  - Laurelton Heart Specialists, Rosedale, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Carl and Edyth Lindner Research Center at The Christ Hospital, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - The Ohio State University College of Medicine, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical School, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University (VCU), Richmond, Virginia
  - University of Washington, Seattle, Washington
  - University of Wisconsin - Madison, Madison, Wisconsin
  - Froedtert & Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (2):
  - Instituto Cardiovascular de Buenos Aires, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Italiano de Buenos Aires, Ciudad Autónoma de Buenos Aires, Buenos Aires
- Australia (8):
  - Liverpool Hospital, Liverpool, New South Wales
  - The Westmead Institute for Medical Research, Westmead, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Advara Heartcare, Leabrook, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Box Hill Hospital, Box Hill, Victoria
  - Advara HeartCare, Joondalup, Western Australia
  - Advara HeartCare Murdoch, Murdoch, Western Australia
- Austria (3):
  - Medizinische Universität Graz, Graz, Styria
  - Medizinische Universität Innsbruck, Innsbruck, Tyrol
  - Medizinische Universität Wien, Vienna
- Belgium (2):
  - Ziekenhuis Oost-Limburg - Campus Sint-Jan, Genk, Limburg
  - Algemeen Ziekenhuis Sint-Jan Brugge-Oostende - Campus Sint-Jan, Bruges, West-Vlaanderen
- Brazil (7):
  - Universidade Estadual de Campinas, Campinas
  - Hospital Moinhos de Vento, Porto Alegre
  - Centro Avançado de Pesquisa e Estudos para o Diagnóstico CAPED, Ribeirão Preto
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto, Ribeirão Preto
  - A Beneficência Portuguesa de São Paulo - Unidade Mirante, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, São Paulo
  - Instituto do Coração de São Paulo, São Paulo
- Canada (6):
  - University of Calgary, Calgary, Alberta
  - Gordon and Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - University Hospital - London Health Sciences Centre, London, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Hôpital Regional de Rimouski, Rimouski, Quebec
- Czechia (3):
  - Fakultní Nemocnice u sv. Anny v Brn, Brno, South Moravian
  - Vseobecna Fakultni Nemocnice v Praze, Prague
  - Institut Klinické a Experimentální Medicíny, Prague
- Denmark (2):
  - Rigshospitalet, Copenhagen, Capital Region
  - Odense Universitetshospital, Odense, Region Syddanmark
- France (6):
  - Hôpital Rangueil, Toulouse, Occitanie
  - Hôpitaux Universitaires Henri Mondor, Créteil
  - Centre Hospitalier Départemental Vendée, La Roche-sur-Yon
  - Hôpital de la Timone, Marseille
  - Hôpital Haut-Lévêque, Pessac
  - Centre Hospitalier Universitaire De Nantes - Hôpital Nord Laennec, Saint-Herblain
- Germany (7):
  - Universitätsklinikum des Saarlandes, Homburg, Saarland
  - Charité Campus Mitte, Berlin
  - Charité Universitätsmedizin Berlin, Berlin
  - Uniklinik Koln, Cologne
  - Universitaetsklinikum Heidelberg - Zentrum fur Innere Medizin, Heidelberg
  - Universitätsklinikum Münster, Münster
  - Universitätsklinikum Würzburg, Würzburg
- Alexandra General Hospital, Athens, Greece
- Israel (3):
  - Rambam Health Care Campus, Haifa
  - Hadassah University Hospital Ein Kerem, Jerusalem
  - Kaplan Medical Center, Rehovot
- Italy (7):
  - Azienda Ospedaliero Universitaria Delle Marche, Ancona
  - Azienda Ospedaliero-Universitaria di Bologna Policlinico Sant Orsola-Malpighi, Bologna
  - Azienda Ospedaliero - Universitaria Careggi, Florence
  - Azienda Ospedale - Università di Padova, Padua
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Fondazione Toscana Gabriele Monasterio per la Ricerca Medica e di Sanita Pubblica, Pisa
  - Azienda Ospedaliera - Universitaria Sant' Andrea, Roma
- Japan (13):
  - Uwajima City Hospital, Uwajima-shi, Ehime
  - Hospital of the University of Occupational and Environmental Health, Kitakyushu-shi, Fukuoka
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Saiseikai Fukuoka General Hospital, Fukuoka, Hukuoka
  - Kokura Memorial Hospital, Kitakyushu, Hukuoka
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Shinshu University Hospital, Matsumoto, Nagano
  - Okayama University Hospital, Okayama, Okayama-ken
  - Osaka Metropolitan University Hospital, Osaka, Osaka
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Keio University Hospital, Shinjuku-Ku, Tokyo
  - Kumamoto University Hospital, Kumamoto
- Poland (2):
  - Krakowski Szpital Specjalistyczny im. Jana Pawa II, Krakow
  - Narodowy Instytut Kardiologii Stefana kardyna Wyszyskiego - Pastwowy Instytut Badawczy, Warsaw
- Portugal (4):
  - Hospital da Senhora da Oliveira - Guimarães, Guimarães
  - Centro Hospitalar Universitário de Lisboa Central - Hospital de Santa Marta, Lisbon
  - Centro Hospitalar Universitário do Porto - Hospital Geral de Santo Antonio, Porto
  - Centro Hospitalar Universitário de São João, Porto
- Veterans Affairs Caribbean Healthcare System, San Juan, Puerto Rico
- Spain (4):
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Skellefteå lasarett, Skellefteå
- United Kingdom (8):
  - Synexus - Scotland Clinical Research Centre, Glasgow, Scotland
  - Synexus - Wales, Cardiff, Wales
  - Synexus Midlands Clinical Research Centre, Edgbaston
  - Synexus - North Tees Clinical Research Centre, Hexham
  - Synexus - Manchester Clinical Research Centre, Liverpool
  - Synexus - Merseyside Clinical Research Centre, Liverpool
  - Royal Free London NHS Foundation Trust, London
  - Richmond Pharmacology, London

IPD SHARING:
Plan to Share IPD: Yes
Ionis may share anonymized individual participant data, aggregated clinical data, and other types of data that support the results in this study. Data requests from qualified researchers will be considered once all three of the following criteria are met: (1) 12 months from marketing approval of the study drug in both the United States and European Union; (2) 18 months from conclusion of the study; and (3) 6 months from publication of study article. Access would be via a secure environment and is contingent upon approval of a research proposal and entry into an appropriate data use agreement. Requests to access data can be submitted via the website https://vivli.org/ourmember/ionis/.